CLINICAL TRIAL: NCT06223139
Title: Association Between Handgrip Strength and Small Airway Disease in Patients with Stable Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: MTU-EC-IM-0-215/65
Record Dates: First submitted 2024-01-12; First posted 2024-01-25 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease; handgrip strength; small airway disease; airway resistance; correlation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD: COPD patients aged 40 years or older with a post-bronchodilator ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) <0.7.
  Interventions: Diagnostic Test: Handgrip strength

INTERVENTIONS:
Diagnostic Test: Handgrip strength — Handgrip strength will be measured by 3 efforts.

SUMMARY:
The goal of this observational study is to investigate the correlation between handgrip strength and small airway disease among patients with chronic obstructive pulmonary disease (COPD). The main question it aims to answer is:

• Is handgrip strength correlated with small airway disease in COPD patients? Participants will perform handgrip strength test and impulse oscillometry (IOS).

DETAILED DESCRIPTION:
This is a cross-sectional study in COPD patients. COPD patients aged 40 years or older were included. Handgrip strength test and impulse oscillometry will be tested in each patient. Handgrip strength will be measured using a hand dynamometer. Small airway disease will be assessed using IOS.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients aged 40 years or older
* Confirmed diagnosis by spirometry (post-bronchodilator FEV1/FVC <0.7)
* Smoking history 10 pack-years or more

Exclusion Criteria:

* COPD exacerbation within 3 months
* Inability to perform handgrip strength test or impulse oscillometry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients aged 40 years or older who are confirmed diagnosis by spirometry (post-bronchodilator FEV1/FVC <0.7) and smoking history 10 pack-years or more.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation between handgrip strength and small airway disease in COPD patients | At day 1 of the study
  This correlation will be reported as correlation coefficient (R).

SECONDARY OUTCOMES:
The best cutoff value of handgrip strength for predicting small airway disease in COPD patients | At day1 of the study
  The best cutoff value will be determined by the area under the Receiver Operator Characteristic curve (ROC).

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Thammasat University Faculty of Medicine, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Keawon T, Saiphoklang N. Association between handgrip strength and small airway disease in patients with stable chronic obstructive pulmonary disease. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241281675. doi: 10.1177/17534666241281675. PMID 39367749